CLINICAL TRIAL: NCT05410145
Title: A Phase 1/2, Open Label, Dose-escalation, and Dose-expansion Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of D3S-001 Monotherapy or Combination Therapy in Subjects With Advanced Solid Tumors With a KRAS p.G12C Mutation
Brief Title: A Study of D3S-001 Monotherapy or Combination Therapy in Subjects With Advanced Solid Tumors With a KRAS p.G12C Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: D3 Bio (Wuxi) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D3S-001-100; 2023-508517-16 (EudraCT Number)
Record Dates: First submitted 2022-05-25; First posted 2022-06-08 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: KRAS P.G12C
Keywords: KRAS p.G12C; Mutation; advanced solid tumors
MeSH Terms: interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- D3S-001 monotherapy (Experimental): Part 1: Dose Escalation, D3S-001 administered orally.
  Part 2 and Part 3a Arm C: Dose Expansion, D3S-001 administered orally in selected cancer type patients.
  Part 4a: Dose Optimization, D3S-001 administered orally in selected cancer type patients.
  Interventions: Drug: D3S-001
- D3S-001 and pembrolizumab (Experimental): Part 3a Arm A: Dose Expansion, D3S-001 in combination therapy administered orally in selected cancer type patients.
  Pembrolizumab administered intravenously.
  Interventions: Drug: D3S-001; Drug: Pembrolizumab
- D3S-001 and platinum doublet chemotherapy (cisplatin + pemetrexed or carboplatin + pemetrexed) (Experimental): Part 3a Arm B: Dose Expansion, D3S-001 in combination therapy administered orally in selected cancer type patients.
  Cisplatin + pemetrexed administered intravenously
  or
  Carboplatin + pemetrexed administered intravenously
  Interventions: Drug: D3S-001; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed
- D3S-001 and Cetuximab (Experimental): Part 3b: Dose Expansion, D3S-001 in combination therapy administered orally in selected cancer type patients.
  Cetuximab administered intravenously.
  Interventions: Drug: D3S-001; Drug: Cetuximab

INTERVENTIONS:
Drug: D3S-001 — Oral
Drug: Pembrolizumab — Intravenous
  Arms: D3S-001 and pembrolizumab
Drug: Cisplatin — Intravenous
  Arms: D3S-001 and platinum doublet chemotherapy (cisplatin + pemetrexed or carboplatin + pemetrexed)
Drug: Carboplatin — Intravenous
  Arms: D3S-001 and platinum doublet chemotherapy (cisplatin + pemetrexed or carboplatin + pemetrexed)
Drug: Pemetrexed — Intravenous
  Arms: D3S-001 and platinum doublet chemotherapy (cisplatin + pemetrexed or carboplatin + pemetrexed)
Drug: Cetuximab — Intravenous
  Arms: D3S-001 and Cetuximab

SUMMARY:
This is a first-in-human (FIH), multicenter, open-label, dose-escalation, and dose-expansion Phase 1/2 clinical trial to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of D3S-001 or combination therapy in subjects with advanced KRAS p.G12C mutant solid tumors. D3S-001 will be taken daily by oral administration in 21-day treatment cycles.

ELIGIBILITY:
Inclusion:

* Subject must have a histologically or cytologically confirmed metastatic or locally advanced solid tumor which is progressing.
* Subject must have documented KRAS p.G12C mutation identified within the last 5 years by a local test on tumor tissue or blood.
* Subject must have measurable disease per RECIST v1.1.
* Subject must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subject must have adequate organ and marrow function within the screening period.

Exclusion:

* Subject has any prior treatment with other treatments without adequate washout periods as defined in the protocol.
* Subject has uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, uncontrolled or significant cardiovascular disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirements, substantially increase risk of incurring AEs, or compromise the ability of the subject to give written informed consent.
* Subject has unresolved treatment-related toxicities from previous anticancer therapy of NCI CTCAE Grade ≥2 (with exception of vitiligo or alopecia).
* Subject has active gastrointestinal disease or other that could interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy.
* Concurrent participation in any clinical research study involving treatment with any investigational drug, radiotherapy, or surgery, except for the nontreatment phases of these studies (e.g., follow-up phase).

Other protocol inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From first dose until 30 days after the last dose (or specified in the protocol).
Number of Participants With Dose-Limiting Toxicities (DLTs) | From Cycle 1 Day 1 through Day 21. Each cycle is 21 days.

SECONDARY OUTCOMES:
D3S-001 maximum observed plasma concentration (Cmax) | Up to 24 months.
D3S-001 time to maximum plasma concentration (tmax) | Up to 24 months.
D3S-001 half-life (t1/2) | Up to 24 months.
D3S-001 area under the concentration-time curve (AUC) | Up to 24 months.
Objective response rate (ORR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Up to 24 months.
Duration of Response (DOR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Up to 24 months.
Progression-free survival (PFS) as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Up to 24 months.
Disease Control Rate (DCR) as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) | Up to 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Chen, MD, Study Director — D3 Bio (Wuxi) Co., Ltd
Locations (51):
- United States (7):
  - D3 Bio Investigative Site 0402, Orange, California
  - D3 Bio Investigative Site 0407, Palo Alto, California
  - D3 Bio Investigative Site 0404, Denver, Colorado
  - D3 Bio Investigative Site 0406, Sarasota, Florida
  - D3 Bio Investigative Site 0401, Detroit, Michigan
  - D3 Bio Investigative Site 0405, Nashville, Tennessee
  - D3 Bio Investigative Site 0403, Houston, Texas
- Australia (5):
  - D3 Bio Investigative Site 0102, Sydney, New South Wales
  - D3 Bio Investigative Site 0101, Malvern, Victoria
  - D3 Bio Investigative Site 0105, Melbourne, Victoria
  - D3 Bio Investigative Site 0103, Nedlands, Western Australia
  - D3 Bio Investigative Site 0104, Bedford Park
- China (16):
  - D3 Bio Investigative Site 0303, Beijing, Beijing Municipality
  - D3 Bio Investigative Site 0306, Guangzhou, Guangdong
  - D3 Bio Investigative Site 0305, Hangzhou, Hangzhou
  - D3 Bio Investigative Site 0307, Harbin, Heilongjiang
  - D3 Bio Investigative Site 0309, Wuhan, Hubei
  - D3 Bio Investigative Site 0312, Wuhan, Hubei
  - D3 Bio Investigative Site 0304, Nanchang, Jiangxi
  - D3 Bio Investigative Site 0302, Shenyang, Liaoning
  - D3 Bio Investigative Site 0310, Jinan, Shandong
  - D3 Bio Investigative Site 0301, Shanghai, Shanghai Municipality
  - D3 Bio Investigative Site 0308, Shanghai, Shanghai Municipality
  - D3 Bio Investigative Site 0316, Chengdu, Sichuan
  - D3 Bio Investigative Site 0311, Hangzhou, Zhejiang
  - D3 Bio Investigative Site 0315, Changsha
  - D3 Bio Investigative Site 0314, Hefei
  - D3 Bio Investigative Site 0313, Zhengzhou
- France (4):
  - D3 Bio Investigative Site 0804, Bordeaux
  - D3 Bio Investigative Site 0803, Lyon
  - D3 Bio Investigative Site 0801, Rennes
  - D3 Bio Investigative Site 0802, Villejuif
- D3 Bio Investigative Site 1002, Hamburg, Germany
- D3 Bio Investigative Site 0501, Shatin, Hong Kong
- Italy (5):
  - D3 Bio Investigative Site 0905, Candiolo
  - D3 Bio Investigative Site 0902, Milan
  - D3 Bio Investigative Site 0904, Napoli
  - D3 Bio Investigative Site 0901, Rome
  - D3 Bio Investigative Site 0903, Siena
- Japan (2):
  - D3 Bio Investigative Site 0601, Kashiwa
  - D3 Bio Investigative Site 0602, Tokyo
- South Korea (4):
  - D3 Bio Investigative Site 0204, Cheongju-si, North Chungcheong
  - D3 Bio Investigative Site 0202, Seoul
  - D3 Bio Investigative Site 0203, Seoul
  - D3 Bio Investigative Site 0201, Seoul
- Spain (6):
  - D3 Bio Investigative Site 0706, Barcelona
  - D3 Bio Investigative Site 0701, Barcelona
  - D3 Bio Investigative Site 0704, Madrid
  - D3 Bio Investigative Site 0705, Madrid
  - D3 Bio Investigative Site 0703, Valencia
  - D3 Bio Investigative Site 0702, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho BC, Lu S, Lee MA, Song Z, Park JJ, Lim SM, Li Z, Zhao J, Richardson G, Zhang Y, Zhang J, Liu A, Loong HH, Chen C, Wang J, Shen Y, Fan Z, Chen Q, Wang H, Zhang J, Chen ZJ, Johnson ML, Mok T. D3S-001 in advanced solid tumors with KRASG12C mutations: a phase 1 trial. Nat Med. 2025 Aug;31(8):2768-2777. doi: 10.1038/s41591-025-03688-6. Epub 2025 Apr 29. PMID 40301557